CLINICAL TRIAL: NCT07327645
Title: The Effect of Proprioceptive Neuromuscular Facilitation on Trunk Mobility, Gait, Fear of Falling, and Quality of Life in Individuals Diagnosed With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Dudu ŞİMŞEK, MSc Physiotherapist, PhD Student,Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PamukkaleU-sımsek-DR-Tez-003
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: PARKINSON DISEASE (Disorder); Proprioceptive Neuromuscular Facilitation; Fear of Falling; Gait Performance; Functional Abilities; Trunk Mobility
Keywords: Proprioceptive neuromuscular facilitation; parkinson disease; trunk mobility; Functional abilities; fear of falling; gait
MeSH Terms: conditions — Parkinson Disease | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Following a power analysis based on the reference study, a total of 42 individuals with PD were included in the study. Randomized according to age, gender, and Hoehn-Yahr level, the individuals were divided into three study groups. While all groups received PNF treatment, Group 1 performed PNF application with physical contact by the physiotherapist, Group 2 with metronome accompaniment, and Group 3 through action observation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with PD-PNF-1 (Experimental): PNF-physiotherapist hand contact group
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF)
- Patients with PD-PNF-2 (Experimental): PNF-Metronom group
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF)
- Patients with PD-PNF-3 (Experimental): PNF-Action Observation Group
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF)

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation (PNF) — Group 2 Treatment Program Warm-up exercises combined with breathing Scapula and pelvis PNF patterns Application of the D2 diagonal in the upper extremity and the D1 diagonal in the lower extremity with slow, opposing technique, without physiotherapist hand contact, accompanied by a metronome Cool-down exercises combined with breathing
  Arms: Patients with PD-PNF-2
Other: Proprioceptive Neuromuscular Facilitation (PNF) — Group 1 Treatment Program Warm-up exercises combined with breathing Scapula and pelvis PNF patterns Application of the D2 diagonal in the upper extremity and the D1 diagonal in the lower extremity with slow, opposing technique, accompanied by physiotherapist's hand contact Cool-down exercises combined with breathing
  Arms: Patients with PD-PNF-1
Other: Proprioceptive Neuromuscular Facilitation (PNF) — Group 3 Treatment Program Warm-up exercises combined with breathing Scapula and pelvis PNF patterns Application of the D2 diagonal in the upper extremity and the D1 diagonal in the lower extremity with slow, opposing technique, under physiotherapist observation, without physiotherapist contact or metronome Cool-down exercises combined with breathing
  Arms: Patients with PD-PNF-3

SUMMARY:
Parkinson's disease (PD) is a neurological disease that includes four main findings: resting tremor, bradykinesia, postural instability, and rigidity, in addition to many motor and non-motor symptoms . PD, the most common form of Parkinsonism, is a chronic and progressive disease characterized by the loss of dopaminergic neurons located in the pars compacta region of the substantia nigra. Its degenerative prognosis, characterized by motor and non-motor problems such as bradykinesia, tremor, rigidity, abnormal postural control, gait disorders, depression, and cognitive impairment, makes the management of the disease difficult . The incidence of PD, which typically begins around the ages of 55-60, varies between 15-250/100,000. Studies conducted in Turkey have indicated an incidence of 202/100,000 . In PH, as the disease progresses, there is a decrease in trunk mobility, forward flexion posture, and consequently loss of postural stability, particularly due to axial rigidity. Trunk stiffness and decreased trunk muscle strength are greater in individuals with PH compared to healthy controls. It has been noted that the decrease in trunk mobility impairs both anterior-posterior and lateral balance, and that individuals with PH experiencing these symptoms have difficulty in timing and scaling effective corrective movements, resulting in an increased risk of falls.

Gait disorders are considered one of the most disabling aspects of PH and can strongly affect the patient's independence and quality of life. The underlying mechanisms of gait disorders are multifactorial and usually result from a multisystem lesion involving both dopaminergic and non-dopaminergic mechanisms . In addition to the clinical and functional effects of gait disorders, a more important issue is that this impairment in gait can result in falls and trauma. The fact that gait disorders are affected by the motor and non-motor symptoms of the disease, and that they are parallel to longevity and cognitive decline, increases the importance of treatment . Therefore, rehabilitation interventions aimed at treating or alleviating gait disorders should be one of the main focuses in individuals with PH .

Falls are one of the most important causes of morbidity for PH . Approximately 60% of PH patients fall at least once a year, and falls are recurrent in at least one-third of these patients . Falls, which occur as a result of various factors, lead to injuries, fear of falling, decreased independence, decreased quality of life, and increased healthcare costs in patients. Fear of falling leads to a decrease in the patient's self-confidence, withdrawal from social life, and the choice of an inactive lifestyle, resulting in an increased risk of falling. This situation becomes a vicious cycle over time. While 28-55% of elderly people living at home fear falling, this rate increases to 50-65% in those who have fallen before . In PH patients, this rate is much higher than in healthy controls and is important in predicting future falls . Therefore, it is stated that fear of falling should be included in the assessment and treatment programs of individuals with PH .

Quality of life is a multidimensional outcome measure consisting of three areas: physical, mental, and social, which are influenced by the individual's personal characteristics and environmental factors . Since chronic and progressive diseases affect every aspect of an individual's life, health-related quality of life is taken into consideration in the management of such diseases . PH affects the individual's ability to independently perform almost all daily living activities and causes negative consequences in quality of life. PH affects the individual not only physically, mentally, and socially, but also economically for the individual and their family due to the additional financial burden brought about by care and treatment costs . Therefore, the assessment of quality of life in individuals with PH is important and necessary .

Proprioceptive Neuromuscular Facilitation (PNF) is a method frequently used by physiotherapists to facilitate the emergence of motor responses through the stimulation of proprioceptors and to improve voluntary control in the central nervous system . The International PNF Association defines the PNF philosophy under 5 subheadings: positive approach (mental participation in therapy), functional approach (integrating real tasks from daily life), mobilizing reserves (radiation principle), holistic treatment of the individual, motor learning, and control principles using motor learning. PNF fully complies with the International Classification of Functioning, Disability and Health (ICF) because it addresses the relevant patient with their personal and environmental context components of deficiencies, activity limitations, and participation restrictions .

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurological disease that includes four main findings: resting tremor, bradykinesia, postural instability, and rigidity, in addition to many motor and non-motor symptoms . PD, the most common form of Parkinsonism, is a chronic and progressive disease characterized by the loss of dopaminergic neurons located in the pars compacta region of the substantia nigra. Its degenerative prognosis, characterized by motor and non-motor problems such as bradykinesia, tremor, rigidity, abnormal postural control, gait disorders, depression, and cognitive impairment, makes the management of the disease difficult . The incidence of PD, which typically begins around the ages of 55-60, varies between 15-250/100,000. Studies conducted in Turkey have indicated an incidence of 202/100,000 . In PH, as the disease progresses, there is a decrease in trunk mobility, forward flexion posture, and consequently loss of postural stability, particularly due to axial rigidity . Trunk stiffness and decreased trunk muscle strength are greater in individuals with PH compared to healthy controls. It has been noted that the decrease in trunk mobility impairs both anterior-posterior and lateral balance, and that individuals with PH experiencing these symptoms have difficulty in timing and scaling effective corrective movements, resulting in an increased risk of falls.

Gait disorders are considered one of the most disabling aspects of PH and can strongly affect the patient's independence and quality of life. The underlying mechanisms of gait disorders are multifactorial and usually result from a multisystem lesion involving both dopaminergic and non-dopaminergic mechanisms. In addition to the clinical and functional effects of gait disorders, a more important issue is that this impairment in gait can result in falls and trauma. The fact that gait disorders are affected by the motor and non-motor symptoms of the disease, and that they are parallel to longevity and cognitive decline, increases the importance of treatment . Therefore, rehabilitation interventions aimed at treating or alleviating gait disorders should be one of the main focuses in individuals with PH .

Falls are one of the most important causes of morbidity for PH . Approximately 60% of PH patients fall at least once a year, and falls are recurrent in at least one-third of these patients . Falls, which occur as a result of various factors, lead to injuries, fear of falling, decreased independence, decreased quality of life, and increased healthcare costs in patients. Fear of falling leads to a decrease in the patient's self-confidence, withdrawal from social life, and the choice of an inactive lifestyle, resulting in an increased risk of falling. This situation becomes a vicious cycle over time. While 28-55% of elderly people living at home fear falling, this rate increases to 50-65% in those who have fallen before . In PH patients, this rate is much higher than in healthy controls and is important in predicting future falls . Therefore, it is stated that fear of falling should be included in the assessment and treatment programs of individuals with PH.Quality of life is a multidimensional outcome measure consisting of three areas: physical, mental, and social, influenced by an individual's personal characteristics and environmental factors . Since chronic and progressive diseases affect every aspect of an individual's life, health-related quality of life is considered in the management of such diseases . PH affects an individual's ability to independently perform almost all daily living activities and leads to negative consequences in quality of life. PH affects the individual not only physically, mentally, and socially, but also economically for the individual and their family due to the additional financial burden of care and treatment costs . Therefore, evaluating the quality of life in individuals with PH is important and necessary.

Proprioceptive Neuromuscular Facilitation (PNF) is a method frequently used by physiotherapists to facilitate the emergence of a motor response through the stimulation of proprioceptors and to improve voluntary control in the central nervous system . The International PNF Association defines the PNF philosophy under 5 subheadings: positive approach (mental engagement in therapy), functional approach (integrating real tasks from daily life), mobilizing reserves (radiation principle), holistic treatment of the individual, motor learning, and control principles using motor learning. PNF fully complies with the International Classification of Functioning, Disability and Health (ICF) because it addresses the relevant patient along with their personal and environmental context components of deficiencies, activity limitations, and participation restrictions.Movements in the human body occur in oblique and rotational directions. In PNF, movements occur as a whole, rotationally and diagonally, and this common direction of movement is called a pattern. Applying PNF exercises in a patterned manner increases the effectiveness of the treatment . In PH, PNF can help individuals achieve efficient motor function and promote benefits related to physical aspects such as clinical condition, tremor, rigidity, bradykinesia, and balance disorders. Theoretical mechanisms for the effect of PNF include autogenic inhibition, reciprocal inhibition, and stress relaxation. These mechanisms could be used to treat rigidity and improve trunk mobility in PH, but there are very few studies reporting them in PH .

A meta-analysis examining PNF applications in individuals with PH included 6 studies. In these studies, PNF application was generally performed in combination with other methods (treadmill training, vibration, gait training), and the patterns were not applied in their pure form . This made it difficult to evaluate the effectiveness of PNF in isolation in individuals with PH. Furthermore, PNF applications in individuals with PH mostly involved lower extremity and pelvic patterns, often focusing on their effects on balance and gait parameters . However, the investigators anticipate that the combined use of upper and lower extremity patterns will have a positive effect on both trunk and gait and balance parameters, and the investigators believe that the PNF technique should be applied to the patient as a single exercise to determine its net effect in PH. The study's findings will contribute to determining the effectiveness of PNF in PH without the need for any additional methods or equipment, thus showcasing its applicability. Furthermore, a review of the literature reveals no studies examining the effects of PNF on trunk mobility, fear of falling, and quality of life. For all these reasons, the investigators believe that this planned study will both fill the gap in the literature and shed light on the treatment of PH patients for physiotherapists working in this field.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease

  * Agreement to participate in the study
  * Age between 40-90 years
  * Score of 21 or higher on the Montreal Cognitive Assessment Scale (MoCA)
  * Hoehn-Yahr stage 1-3 (including 3)

Exclusion Criteria:

* • Refusal to participate in the study

  * Having vision loss (can wear glasses or contact lenses)
  * Having hearing loss (can wear a hearing aid)
  * Being in Hoehn-Yahr stage 4-5
  * Having accompanying neurological, orthopedic, and rheumatological diseases that prevent the performance of upper and lower extremity patterns.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
The Modified Hoehn and Yahr Scale | 10 weeks after the start of treatment
  Parkinson's Hoehn and Yahr Staging is a scale developed in 1967 by Margaret M. Hoehn and Melvin D. Yahr that examines the overall clinical condition of individuals with Parkinson's disease according to five stages. Advanced stage indicates an increased stage. It provides information about objective findings and functional impairment of the disease. Although initially designed as a 5-item scale with integer options from 1 to 5, some items with 0.5-point increments were later added.

SECONDARY OUTCOMES:
The Movement Disorders Association-Unified Parkinson's Disease Rating Scale (MDS-UPRDS | 10 weeks after the start of treatment
  The Movement Disorders Association-Unified Parkinson's Disease Rating Scale (MDS-UPRDS) is the most widely used of all clinical scales currently available for assessing motor impairment and disability in PD. The scale results in a score indicating the severity of the disease (35). It evaluates motor performance, mental and emotional status, and activities of daily living. In addition to these, the scale also assesses motor fluctuations, dyskinesias, and autonomic dysfunction that may occur as complications of levodopa treatment (36). The first section consists of 4 questions, the second section 13, and the third section 14. The fourth section is divided into three subsections (A-B-C). Sections A and B consist of 4 questions each, and section C consists of 3 questions. The higher the score, the greater the severity of the disease in PD.
Parkinson's Disease Questionnaire (PDQ-39): | 10 weeks after the start of treatment
  Parkinson's Disease Questionnaire (PDQ-39): It is a valid, reliable and sensitive scale widely used to assess quality of life in individuals with PD. It consists of 39 questions in total, with sub-parameters including mobility, activity of daily living, emotional well-being, stigma, social support, cognition, communication and physical discomfort. The total score obtained from the scale ranges from 0 to 100. As the score increases, the quality of life deteriorates (37). A Turkish validity and reliability study of PHA-39 has been conducted.
Modified Fall Activity Scale (MFES): | 10 weeks after the start of treatment
  Modified Fall Activity Scale (MFES): The Fall Activity Scale (FES) is the most widely used and best-known questionnaire for measuring fall-related confidence. The MFES aims to measure a person's perceived confidence while performing 10 defined daily living activities. The MFES is an expanded version developed by Hill et al., incorporating four additional outdoor activity tasks. With good scaling properties and test-retest reliability, the MFES is a clear and simple tool consisting of 14 questions used to assess fear of falling, scoring the activity in question on a scale of 0-10. The Turkish validity and reliability of the scale were established by Korkmaz et al.
Modified Schober test | 10 weeks after the start of treatment
  This test was first described in 1937 by the German physician Paul Schober, and the method was modified by Macrae and Wright in 1969. In this test, while the person is in an upright position, the lumbosacral junction and 10 cm above it are marked. Then, a third mark is placed 5 cm below the lumbosacral junction. After anterior flexion performed as far forward as possible, the distance between the highest and lowest marks is measured with a tape measure or inclinometer. A distance of 4 cm or less indicates restricted lumbar movement. The modified Schober test is used in the assessment of spinal mobility.
Timed Up and Go Test (TUG) | 10 weeks after the start of treatment
  The TUG, which includes walking and turning functions, has been shown to be highly reliable and valid for individuals with PH (28,29). It can accurately identify individuals with PH at risk of falling with 74% accuracy (43). The person undergoing the test sits in a chair of normal height. Upon the command "Start," the person is asked to stand up from the chair, walk 3 meters forward at a normal walking speed, and then return and sit back in the chair (43). It is generally administered twice, and the average time is recorded. The person is allowed to use an assistive device (if any), and this is noted (44). A time ≤10 seconds indicates that the patient walks independently and has a low risk of falling; a time >30 seconds indicates that the patient occasionally needs assistance and has a high risk of falling (45). The TUG will first be administered in isolation, and then repeated with a cognitive task (counting backward from 100 in increments of 3).
Spatio-Temporal Gait Analysis: | 10 weeks after the start of treatment
  Gait analysis is the evaluation of neuromusculoskeletal system functions and the interpretation of results using numbers and graphs. While gait analysis can be performed visually, the human eye is insufficient to perceive movements within milliseconds, necessitating measurement with technological devices. Gait analysis devices make it possible to measure and evaluate force, moment, and muscle activity. Thanks to these systems, all stages of walking can be recorded completely, converted into numerical data, before/after comparisons can be made, and changes can be evaluated.
Statistical Analysis | 10 weeks after the start of treatment
  Data were analyzed using SPSS 22.0 [IBM SPSS Statistics 22 software ® (Armonk, NY: IBM Corp.)]. Continuous variables were presented as mean ± standard deviation, median, and 25-75% interquartile range, while categorical variables were presented as number (n) and percentage (%). Differences between categorical variables were examined using Chi-Square analysis. Since parametric test assumptions were not met, the Wilcoxon signed-rank test was used to compare differences in the dependent group. The Kruskal-Wallis H test was used to compare differences in the independent group. The Mann-Whitney U test was used for pairwise comparisons of independent groups. Since there was more than one independent variable, partial eta-squared (partial η2) was used to calculate the effect strength of the independent variable on the dependent variable, controlling for the main and joint effects of other independent variables. A partial η2 value of 0.01 indicated low effect strength, 0.06 indicated average

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale Unıversity, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alexandre de Assis IS, Luvizutto GJ, Bruno ACM, Sande de Souza LAP. The Proprioceptive Neuromuscular Facilitation Concept in Parkinson Disease: A Systematic Review and Meta-Analysis. J Chiropr Med. 2020 Sep;19(3):181-187. doi: 10.1016/j.jcm.2020.07.003. Epub 2020 Dec 15. PMID 33362441